CLINICAL TRIAL: NCT04343638
Title: Effect of Intraoperative Nociception Control Based on Analgesia Nociception Index (ANI) Monitoring on Stress Response During Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2020-0130
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Patients Undergoing Total Laparoscopic Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will be randomly allocated to 2 groups using computer-generated randomization method. Anesthesiologists will not be blinded to the groups because of organizational reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional nociception control arm (Active Comparator): Intraoperative opioid will be administered by conventional clinical practice. ANI monitor readings will not be visible to the anesthesiologist.
  Interventions: Device: conventional nociception control
- ANI-monitor guided nociception control arm (Experimental): Intraoperative opioid will be administered by maintaining the 4-minute moving average of ANI ≥50.
  Interventions: Device: ANI monitor guided nociception control

INTERVENTIONS:
Device: conventional nociception control — While Intraoperative opioid will be administered by conventional clinical practice in control arm.
  Arms: conventional nociception control arm
Device: ANI monitor guided nociception control — The intraoperative opioid will be administered by maintaining the 4-minute moving average of ANI ≥50 in ANI-monitor guided nociception control arm.
  Arms: ANI-monitor guided nociception control arm

SUMMARY:
The "Analgesia Nociception Index" (ANI; MetroDoloris Medical Systems, Lille, France), derived from an electrocardiogram (ECG) trace, has been proposed as a noninvasive guide to analgesia. The ANI monitor calculates HR variation with respiration, a response mediated primarily by changes in the parasympathetic nervous system (PNS) stimulation to the sinoatrial node of the heart. The aim of this study is to determine the relation between ANI monitor values and serum catecholamine levels. We will compare the serum catecholamine (norepinephrine, epinephrine) levels of conventional nociception control group and ANI-monitor guided nociception control group at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing total laparoscopic hysterectomy under general anesthesia (American society of anesthesiologists classification 1~3)

Exclusion Criteria:

1. endometriosis
2. AP diameter of uterus > 12cm
3. cognitive disorder
4. arrhythmia, pacemaker
5. chronic opioid use
6. diseases affecting autoimmune system (immune disease, diabetic neuropathy)
7. use of medications affecting ANI monitor (antimuscarinics, alpha-agonist, beta blocker)
8. illiteracy, foreigner

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Serum catecholamine (norepinephrine, epinephrine) level at the end of surgery | at the end of surgery (skin closure)
  Blood samples for serum catecholamine (norepinephrine, epinephrine) will be drawn at the end of surgery and 1 hour after the end of surgery..

SECONDARY OUTCOMES:
plasma inflammatory markers (IL-6, IL-10, HMGB1) | at the end of surgery (skin closure) and 1 hour after the end of surgery
  Blood samples for plasma inflammatory markers (IL-6, IL-10, HMGB1) will be drawn at the end of surgery (skin closure) and 1 hour after the end of surgery.
hormone level (cortisol, adrenocorticotropic hormone) | at the end of surgery (skin closure) and 1 hour after the end of surgery
  blood samples for hormone levels (cortisol, adrenocorticotropic hormone) will be drawn at the end of surgery (skin closure) and 1 hour after the end of surgery.
serum catecholamine (norepinephrine, epinephrine) level | 1 hour after the surgery
  Blood samples for serum catecholamine (norepinephrine, epinephrine) will be drawn 1hour after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Chang CH, Lee JR, Seo SK, Kwon YI, Lee JH. Effect of analgesia nociception index monitor-based nociception control on perioperative stress responses during laparoscopic surgery in Trendelenburg position: a randomized controlled trial. Front Med (Lausanne). 2023 Aug 4;10:1196153. doi: 10.3389/fmed.2023.1196153. eCollection 2023. PMID 37601786